CLINICAL TRIAL: NCT03401359
Title: Prospective Longitudinal Biomarker Study of Acquired Resistance and Immune Response to Palbociclib in Breast Cancer
Brief Title: The Resistance and Immune Response to Palbociclib in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-07-049
Record Dates: First submitted 2017-12-11; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: tissue biopsy, blood sample — At baseline, 100 tumor/blood samples will be banked. Only ~60 will be profiled if the paired samples are acquired post-progression or on-treatment. On-treatment blood samples will be serially collected and banked from all consenting patients.

SUMMARY:
The investigators propose to conduct a biomarker and molecular profiling study in longitudinally paired tumor biopsies and serum from patients with Hormone Receptor positive (HR+) metastatic Breast Cancer (BC) treated with Palbociclib in combination with endocrine therapies.

DETAILED DESCRIPTION:
The investigators propose to conduct a biomarker and molecular profiling study in longitudinally paired tumor biopsies and serum from patients with Hormone Receptor positive (HR+) metastatic Breast Cancer (BC) treated with Palbociclib(Palbo) in combination with endocrine therapies.

The investigators plan to obtain tumor biopsy and blood samples, taken at both pre-treatment and post-progression, from 40 patients who develop acquired resistance to Palbo + endocrine combination treatment. All assays will be conducted in parallel on both pre and post-treatment samples to identify differences that may account for acquired resistance. Cyclin E1 and E2 levels will be assessed by IHC on tumor biopsies. Neuregulin-1 levels will be assessed by ELISA assay on serum. Tumor biopsies will be further profiled using whole-exome sequencing (WES) and whole-transcriptome sequencing (RNA-Seq). Matched blood samples will be subject to WES to facilitate somatic mutation detection. Paired tumor biopsies will undergo immunohistochemistry (IHC) analysis of TIL markers to assess Palbo-induced changes. Finally, we will apply the in-house circulating tumor DNA (ctDNA) assay, which employs a custom-designed panel for studying Palbo acquired resistance, towards the analysis of 40 pairs of plasma samples. The custom ctDNA panel will be extended to include additional mutations identified from this study that confer acquired resistance.

To further evaluate the effects of Palbo treatment on intratumoral TILs, the investigators plan to acquire paired tumor biopsy and matched blood samples, at baseline and two time points (6 weeks, 12 weeks) during the course of Palbo treatment, from 20 patients. And they will select metastatic BC patients who exhibit stable diseases (SD) in response to Palbo for tumor biopsies, prior to knowledge of whether post-progression biopsy would be available. Tumor biopsies will be subject to WES, RNA-Seq and IHC analyses. Further, the investigators plan to quantify the abundance of immune cell sub-populations in the matched blood samples using flow cytometry (FACS) to assess Palbo treatment effects on systematic immunity.

While on-treatment samples can be collected after 6 weeks and 12 weeks of initiating Palbo treatment, it takes about 18 months on average for initially treated patients with late stage HR+ breast cancers to develop acquired resistance. Only an estimated 40% of relapsed cases will have successful biopsies due to a lack of consent or difficult-to-operate biopsies such as bone-only metastases. Hence, the investigators plan to bank pre-treatment biopsies and blood samples from about 100 patients by Q2 2018 in order to collect 40 post-progression biopsies as matched pairs within the 2-year time frame. FFPE slides will be made from all tumor biopsies, including the 100 cases at baseline, and subject to H&E staining. The investigators will detect and quantify TILs through machine learning and digital imaging analysis of the H&E data.

ELIGIBILITY:
Inclusion Criteria:

* Hormone receptor positive, metastatic breast cancer
* Treated by palbociclib with endocrine therapy

Exclusion Criteria:

* Hormone receptor negative breast cancer
* Treated without palbociclib
* Refuse and withdrawal to this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker of palbociclib in metastatic breast cancer | 24.8 months (median progression free survival in palbociclib plus letrozole treatment (according to PALOMA-2 trial)
  Biomarker of acquired resistance and immune response to palbociclib in metastatic breast cancer from whole exome sequencing, RNASeq, circulating tumor DNA and flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park YH, Im SA, Park K, Wen J, Lee KH, Choi YL, Lee WC, Min A, Bonato V, Park S, Ram S, Lee DW, Kim JY, Lee SK, Lee WW, Lee J, Kim M, Kim HS, Weinrich SL, Ryu HS, Kim TY, Dann S, Kim YJ, Fernandez DR, Koh J, Wang S, Park SY, Deng S, Powell E, Ravi RK, Bienkowska J, Rejto PA, Park WY, Kan Z. Longitudinal multi-omics study of palbociclib resistance in HR-positive/HER2-negative metastatic breast cancer. Genome Med. 2023 Jul 20;15(1):55. doi: 10.1186/s13073-023-01201-7. PMID 37475004